CLINICAL TRIAL: NCT00037882
Title: A Phase II Study of SCH 54031 (Peg Interferon Alpha-2B/PEG-Intron) in Subjects With Interferon-Refractory Chronic Myelogenous Leukemia
Brief Title: PEG-Intron For Chronic Myelogenous Leukemia Patients Unresponsive To Or Intolerant Of Roferon Or Intron
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM00-150
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Myeloid, Philadelphia-Positive
Keywords: Chronic Myelogenous Leukemia; Interferon alpha; Roferon; Intron; Chronic Myelogenous Leukemia-Philadelphia positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCH 54031 (Experimental): Peg Interferon Alpha-2B/PEG-Intron
  Interventions: Drug: PEG-Intron

INTERVENTIONS:
Drug: PEG-Intron — Once weekly injection.
  Other Names: SCH 54031; Peg Interferon Alpha-2B

SUMMARY:
The purpose of this study is to determine if PEG-Intron is better tolerated and more efficacious than standard interferons (Roferon, Intron) in patients with Philadelphia-positive Chronic Myelogenous Leukemia. These patients should have previously received standard interferon therapy and have been intolerant, resistant, or have relapsed disease.

DETAILED DESCRIPTION:
It has been shown that patients who experience complete hematologic or at least a partial cytogenetic response to interferon will have improved survival times. In addition, evidence exists that even patients who do not demonstrate a cytogenetic response to interferon treatment can still benefit from treatment, in terms of survival, compared to patients not treated with interferon. This indicates that if a patient is better able to tolerate interferon, he or she may have improved survival even without cytogenetic response. Preliminary studies suggest that PEG-Intron is more convenient for patients (administered once weekly rather than daily), is better tolerated than interferon, and can produce hematologic remission in interferon-a resistant patients. Phase II studies are needed to ascertain the overall hematologic and cytogenetic response rates to PEG-Intron in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic phase CML, documented by the presence of Philadelphia chromosome or bcr/abl rearrangement at time of diagnosis, confirmed by either cytogenetics or PCR.
* WBC >/= 3000/ul </=100,000/ul.
* Patients must have received prior interferon therapy & proven to have primary refractory disease, secondary resistance or intolerance to interferon-a
* Patient must have ECOG status of 0, 1, or 2
* Labs: SGOT/SGPT<2xULN; serum bilirubin<2xULN; serum creatinine <2.0mg/dl
* Recovered from effects of major surgery
* Life expectancy > 12 wks.
* Signed informed consent.
* Women of childbearing potential must have negative serum pregnancy test within 72 hrs prior to administration of PEG-Intron & use effective contraception during the study.

Exclusion Criteria:

* NO accelerated Phase CML patients with peripheral blood: blasts>/=15%, basophils>/=20%, blasts+promyelocytes>/=30%, platelets<100,000/ul (unrelated to therapy). Blastic phase CML:>/=30% in peripheral blood/bone marrow.
* NO patients with known hypersensitivity to interferon-a.
* NO severe cardiovascular disease, i.e. arrhythmias requiring chronic treatment or congestive heart failure (NYHA classification III/IV).
* NO history of neuropsychiatric disorder requiring hospitalization.
* NO patients requiring therapy for refractory thyroid dysfunction
* NO patients with uncontrolled diabetes mellitus.
* NO patients who have had treatment for a 2nd malignancy in the past 5 yrs, except for localized basal cell/squamous cell carcinoma of the skin or cervical carcinoma in situ.
* NO pregnant or lactating patients.
* NO patients known to be actively using alcohol or drugs
* NO patients receiving any experimental therapy within 30 days of enrollment in study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2001-02 (Actual); Primary Completion 2003-12-03 (Actual); Study Completion 2003-12-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, M.D., Study Chair — UT MD Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Public website for M.D.Anderson Cancer Center — http://www.mdanderson.org